CLINICAL TRIAL: NCT03068078
Title: A Reduced-carbohydrate Diet High in Monounsaturated Fats in Type 2 Diabetes: a Six-month Study of Changes in Metabolism, Liver- and Cardiovascular Function (ReDuCtion)
Brief Title: A Reduced-carbohydrate Diet High in Monounsaturated Fats in Type 2 Diabetes
Acronym: ReDuCtion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Danish Diabetes Academy (Other); Region of Southern Denmark (Other); Odense Patient Data Explorative Network (Other); Novo Nordisk A/S (Industry); University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Aleksander Krag, Professor, PhD, M.D., DMSc, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-20150217
Record Dates: First submitted 2017-01-26; First posted 2017-03-01 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-07

CONDITIONS: Type2 Diabetes; Nonalcoholic Steatohepatitis; Non-Alcoholic Fatty Liver Disease; Atherosclerosis; Dyslipidemias
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Atherosclerosis; Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control-group (No Intervention): The control group will be eating a regular diabetes diet according to the Danish National Recommendations
- Intervention-group (Experimental): Intervention-group will be eating a low carbohydrate diet, high in monounsaturated fats
  Interventions: Dietary Supplement: Low carbohydrate diet high in monounsaturated fats

INTERVENTIONS:
Dietary Supplement: Low carbohydrate diet high in monounsaturated fats — Participants will have to change their diet during 6 months
  Other Names: LCD
  Arms: Intervention-group

SUMMARY:
Further studies are needed to establish the optimal diet for treating T2D.

The investigators wishes to investigate whether a low carbohydrate diet, high in monounsaturated fats (LCD) will affect cardiovascular function, metabolism and the liver.

135 participants with T2D, will be following either a LCD, or a regular diabetes diet (RDD) for 6 months. Measurements and investigations will be performed at baseline and after 6 months.

DETAILED DESCRIPTION:
Type 2 diabetes (T2D) is an increasing global problem, especially in developing countries. T2D is associated with an increased risk of cardiovascular disease (CVD), where hyperglycemia is especially important for microvascular damage.

Previous studies in T2D on reduced carbohydrate intake has shown beneficial effects on glycemic control, indicated by reduction in HbA1c, fasting insulin and 2h-glucose (OGTT) values. However further studies are needed to establish the optimal diet for treating T2D.

The investigators wishes to investigate whether a low carbohydrate diet, high in monounsaturated fats will:

1. Improve glycemic control, dyslipidemia and metabolic markers in T2D despite unchanged anti-diabetic treatment.
2. Improve endothelial function assessed by flow-mediated vasodilation (FMD) in the brachial artery as well as microvascular damage assessed by retinal scan, urine albuminuria and minimal forearm vascular resistance (MFVR).
3. Improve Non-Alcoholic Fatty Liver Disease (NAFLD) assessed by >2 points reduction in NAFLD Activity score with at least 1 point reduction in either lobular inflammation or hepatocellular ballooning, without worsening of fibrosis.
4. Improve quality of life
5. Improve gut dysbiosis

The study will be conducted through a 6 month randomized controlled trial with 135 participants with type 2 diabetes. 90 participants will be randomized to the intervention group, following a LCD, and 45 participants will be randomized to the control group (regular diet for diabetes, RDD). The below described measurements will be conducted before baseline and after 6 months, and the participants will fill out a QoL questionnaire at 0, 3 and 6 months.

Planned examinations are ultrasound assessment of flow-mediated vasodilation, Dual-energy X-ray absorptiometry (DEXA-scan), retina scan, liver biopsy, liver-scans, blood, urine, hair, saliva and feces. Accelerometers will be applied before, during and after the study to evaluate compliance in unchanged exercise pattern. Compliance with diet will be evaluated by a clinical dietitian and through food diaries.

Baseline histology from the first 50 participants suggest that the current inclusion criteria doesn't cover the full spectrum of NAFLD (NASH and fibrosis) as expected. Further 50 participants who will have had diabetes for more than 10 years and who will not fulfill inclusion criteria number 1 and 2 will be included. On this group of participants we will only perform liver-investigations and DEXA-scan. This group of participants, will not affect the timeschedule of the main study.

ELIGIBILITY:
Inclusion Criteria:

1. Duration of established T2D for more than six months and less than five years and HbA1c in compliance with T2D (above 48 mmol/mol), but without need for adjustment of antidiabetic treatment*
2. Serum cholesterol below 4.5 mmol/l and LDL cholesterol below 2.5 mmol/l at inclusion**
3. Age of 18 or above
4. Stable diabetic treatment three months prior to inclusion***
5. Be able to read and understand Danish language
6. Signed written consent

   * based on the assumption that metabolic and cardiovascular changes are less likely to be reversible in patients with longstanding T2D. HbA1c and need for adjustment and if the patient is eligible for inclusion will be evaluated individually based on the patients current treatment and current HbA1c by the project responsible. If the patient has duration of diabetes > 5 years but with current treatment ≤ 2 oral antidiabetic drugs and without insulin treatment, the patient will be accepted for enrolment.

     * To avoid changes in lipid-lowering treatment during follow-up total cholesterol should be below 4.5 mmol/l and LDL cholesterol below 2.5 mmol/l at inclusion. Higher levels may be accepted if the patient cannot tolerate lipid-lowering treatment ***Patients can be enrolled three months after medication change

Exclusion Criteria:

1. Low carbohydrate diet prior to inclusion
2. Hypoglycemic unawareness
3. Excessive weight loss within the last three months, defined as more than 10 kilograms
4. Current treatment with glucocorticoids (systemic)
5. Continuous treatment with steatosis-inducing drugs (e.g. carbamazepine)
6. Treatment with antibiotics up to 2 months before inclusion*
7. Treatment with chemotherapy
8. Pregnancy or expected pregnancy within the next 6 months
9. Active alcohol overuse**
10. Active cancer
11. Significant co morbidity including liver disease
12. Poor compliance *Participants can be rescheduled to be included 2 months after use of antibiotics ** Prior alcohol overuse and eligibility will be evaluated individually

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2021-06-04 (Actual)

PRIMARY OUTCOMES:
Glycemic control, dyslipidemia and metabolic markers | Change from baseline at 6 months
  Measured by HbA1c, serum cholesterol, blood glucose and metabolic markers

SECONDARY OUTCOMES:
Endothelial function | Change from baseline at 6 months
  assessed by FMD in the brachial artery as well as microvascular damage assessed by retinal scan, urine albuminuria and minimal forearm vascular resistance (MFVR).
Non-Alcoholic Fatty Liver Disease (NAFLD) | Change from baseline at 6 months
  Assessed by >2 points reduction in NAFLD Activity score with at least 1 point reduction in either lobular inflammation or hepatocellular ballooning, without worsening of fibrosis.
Quality of life | Change from baseline at 6 months
  Assessed by questionaire
Gut dysbiosis | Change from baseline at 6 months
  Assessed by fecal sample

CONTACTS AND LOCATIONS:
Overall Officials: Henning Beck-Nielsen, Professor, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Petersen EE, Hansen JK, Torp N, Gram-Kampmann E, Andersen P, Johansen S, Villesen IF, Bech KT, Thorhauge KH, Schnefeld HL, Bastida Gjol CM, Jensen EL, Detlefsen S, Hojlund K, Thiele M, Israelsen M, Krag A, Hansen CD. Health-related quality of life, compliance and sustained adherence on a Low-Carbohydrate High-Fat diet compared with a High-Carbohydrate Low-Fat diet in people with type 2 diabetes. Am J Clin Nutr. 2026 Jan 27:101211. doi: 10.1016/j.ajcnut.2026.101211. Online ahead of print. PMID 41611090
- [Derived] Wernberg CW, Indira Chandran V, Lauridsen MM, Skytthe MK, Hansen CD, Hansen JK, Gronkjaer LL, Jacobsen BG, Di Caterino T, Detlefsen S, Thiele M, Guiliani AM, Villesen IF, Leeming DJ, Karsdal M, Graversen JH, Krag A. Ability of soluble TREM2 and PRO-C3 as biomarkers to predict changes in MASLD activity. JHEP Rep. 2025 Apr 22;7(8):101432. doi: 10.1016/j.jhepr.2025.101432. eCollection 2025 Aug. PMID 40677693
- [Derived] Gram-Kampmann EM, Olesen TB, Hansen CD, Hugger MB, Jensen JM, Handberg A, Beck-Nielsen H, Krag A, Olsen MH, Hojlund K. A six-month low-carbohydrate diet high in fat does not adversely affect endothelial function or markers of low-grade inflammation in patients with type 2 diabetes: an open-label randomized controlled trial. Cardiovasc Diabetol. 2023 Aug 17;22(1):212. doi: 10.1186/s12933-023-01956-8. PMID 37592243
- [Derived] Hansen CD, Gram-Kampmann EM, Hansen JK, Hugger MB, Madsen BS, Jensen JM, Olesen S, Torp N, Rasmussen DN, Kjaergaard M, Johansen S, Lindvig KP, Andersen P, Thorhauge KH, Brond JC, Hermann P, Beck-Nielsen H, Detlefsen S, Hansen T, Hojlund K, Thiele MS, Israelsen M, Krag A. Effect of Calorie-Unrestricted Low-Carbohydrate, High-Fat Diet Versus High-Carbohydrate, Low-Fat Diet on Type 2 Diabetes and Nonalcoholic Fatty Liver Disease : A Randomized Controlled Trial. Ann Intern Med. 2023 Jan;176(1):10-21. doi: 10.7326/M22-1787. Epub 2022 Dec 13. PMID 36508737